CLINICAL TRIAL: NCT06071429
Title: Bioresorbable Sirolimus-Eluting Scaffold Treatment for Below the Knee Disease
Acronym: ELITE-BTK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: R3 Vascular Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP001
Record Dates: First submitted 2023-09-28; First posted 2023-10-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAGNITUDE BRS (Experimental): Participants who receive the MAGNITUDE BRS device will be included in this arm
  Interventions: Device: MAGNITUDE Sirolimus-eluting Bioresorbable Scaffold
- Percutaneous Transluminal Angioplasty (PTA) (Active Comparator): Participants who receive a PTA device will be included in this arm
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA)

INTERVENTIONS:
Device: MAGNITUDE Sirolimus-eluting Bioresorbable Scaffold — CLTI patients treated with MAGNITUDE BRS
  Arms: MAGNITUDE BRS
Device: Percutaneous Transluminal Angioplasty (PTA) — CLTI patients treated with PTA
  Arms: Percutaneous Transluminal Angioplasty (PTA)

SUMMARY:
The objective of this prospective, single-blinded, randomized controlled trial is to evaluate the safety and efficacy of the MAGNITUDE BRS System for the planned treatment of narrowed infrapopliteal lesions. Approximately 276 subjects will be randomized in a 1:1 ratio. The clinical investigation will be conducted at up to 60 clinical sites globally.

ELIGIBILITY:
General Inclusion Criteria

1. Subject (or their legally authorized representative) has provided written informed consent prior to any study-related procedure, using the form approved by the Institutional Review Board / Ethics Committee.
2. Subject agrees not to participate in any other investigational device or drug study for a period of at least 12 months following the index procedure.

   Note: Questionnaire-based studies, or other studies that are non-invasive and do not require investigational devices or medications are allowed.
3. Subject has symptomatic chronic limb-threatening ischemia, determined as Rutherford categories 4 or 5.
4. Subject is ≥ 18 years of age.
5. Subject agrees to complete all protocol-required follow-up visits, including angiograms.

   Angiographic Inclusion Criteria
6. Target lesion(s) in the infrapopliteal vessel(s) of the same limb located in any of the following vessels: tibioperoneal trunk (TPT), anterior tibial artery (ATA), posterior tibial artery (PTA), or peroneal artery.
7. Target lesion(s) must be located in the proximal 2/3 of the native infrapopliteal vessels and at least 10 cm above the tibio-talar joint.

   Note: Up to two (2) target lesions and two different arteries can be treated
8. All target lesions must be successfully crossed with a guidewire prior to randomization.

   Note: For CTO, retrograde crossing of the lesion is allowed but treatment must be via antegrade.

   Note: The most distal lesion must be treated before treating more proximal lesions.
9. Distal tibial and pedal runoff for each target lesion must be patent (free of lesions with < 50% stenosis). If the index vessel is either anterior or posterior tibial artery, outflow must be contiguous with a patent dorsalis pedis or common plantar artery.
10. Inflow above-the-knee lesions must be treated successfully (< 30% diameter stenosis by angiography without evidence of distal embolization, thrombus formation, or vessel rupture).

    Note: Inflow lesions may be treated during the index procedure prior to target lesion(s) using the standard of care (including drug-eluting devices), without wiring the target lesion, if possible. Treatment of inflow lesions in the target limb within prior 30 days is also allowed provided the treatment was successful.

    Note: Atherectomy of non-target lesions is not allowed.
11. Target lesion must have reference vessel diameter is between 2.75 - 3.75 mm by angiography. Vessel size measured by IVUS is highly recommended to verify RVD.
12. Target lesion(s) is de novo or restenosed ≥ 70% stenosed by angiography. Note: In-stent restenosis is an exclusion criterion.
13. The total target lesion length among all target lesions must not exceed 11 cm.
14. Minimum target lesion length must be >14 mm.
15. Total scaffold length must not exceed 12 cm, and include at least 2 mm of normal vessel from each pre-dilatation border.
16. The target vessel must not have any other angiographic significant non-target lesions (≥ 50%).
17. Tandem non-contiguous target lesions are allowed if there is a plaque-free zone of ≥ 2 cm between the lesions. Total lesion lengths must not exceed 11 cm.
18. Target lesion(s) stenting does not block access to patent main named branches (tibioperoneal trunk (TPT), anterior tibial artery (ATA), posterior tibial artery (PTA), or peroneal artery).
19. Non-target below-the-knee lesions in non-target vessels must be successfully treated per standard of care prior to randomization without evidence of thrombosis, distal embolization, or vessel rupture.

    Note: Drug-eluting and atherectomy devices for treatment of non-target lesions is not allowed.
20. Subject has suitable common femoral (contralateral or antegrade ipsilateral) vascular access.

    Note: Retrograde pedal approach is allowed for crossing but not for treatment of target lesion(s).
21. At least one fully patent below-the-ankle artery (i.e., dorsalis pedis; common with either, lateral, or medial plantar arteries) without hemodynamically significant lesions (≥ 50% diameter stenosis by angiography) must be present in the target limb.

General Exclusion Criteria

Subjects must not meet any of the following general and angiographic exclusion criteria:

1. Subject with Body Mass Index (BMI) < 18.
2. Subject is pregnant or nursing. Subjects who plan pregnancy during the clinical investigation follow-up period may not be enrolled.

   Note: Subjects of child-bearing potential must have a negative pregnancy test ≤ 28 days prior to the index procedure and agree to use contraception for 6 months.
3. Estimated life expectancy <1 year, in the opinion of the Investigator at the time of enrollment.
4. Subject is permanently bedridden.
5. Subject has known hypersensitivity or contraindication to device materials and their degradants (sirolimus, poly (L-lactide), poly (D, L-lactide), lactic acid, or platinum-iridium) or to study medications (including antiplatelet medications) or to contrast media and who cannot be adequately premedicated.
6. Subject has planned surgery or procedure necessitating discontinuation of antiplatelet medications within 6 months after the index procedure.
7. Subject has had revascularization procedure within the target vessel in the previous 3 months
8. Subject has prior major amputation (above or below the knee or above the ankle) involving the target limb.

   Note: Major amputation of the contralateral limb is allowed.
9. Subject has planned surgical or endovascular procedure within 6 months following the index procedure.

   Note: A planned minor amputation (toe and/or transmetatarsal amputation in either limb) is allowed. Treatment of inflow lesions in the target limb within prior 30 days is also allowed provided the treatment was successful (< 30% residual stenosis, no thrombi, distal emboli or vessel rupture).
10. Subject who has severe ischemia (ABI ≥ 0.39).
11. Subject who has neuropathic lesion(s) with no ischemic component (wounds or ulcers occur on pressure zones of the foot with or without Type 2 diabetes , deformed foot/toes, hematoma, edema ).
12. Subject has presence of osteomyelitis or any gangrene above the metatarsal-phalangeal joints, extensive tissue loss with exposed tendons or requiring complex or recurrent surgeries, full thickness heel ulcer, or pure neuropathic ulcers.
13. Subject with uncontrolled diabetes with HbA1c > 10%.
14. Subject has a prior stroke or myocardial infarction within 3 months of the index procedure.
15. Subject has acute renal failure, severe or end-stage chronic kidney disease (eGFR < 30 mL/min), or requires dialysis.
16. Subject has active systemic infection.
17. Subject is receiving immunosuppression therapy and/or has known immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, rheumatoid arthritis, severe asthma requiring immunosuppressive medication, etc.).
18. Subject has active malignancy (receiving or scheduled to receive anticancer therapy for malignancy within 1 year prior to or after the index procedure), active blood dyscrasia or coagulation disorder (platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC < 3,000 cells/mm3, or hemoglobin < 8.0 g/dl).
19. Subject is an incapacitated individual, defined as a person who is mentally ill, mentally handicapped, or an individual without legal authority to control their activities.
20. Subject has significant comorbid condition(s), or other medical, social, or psychological conditions (such as history of substance abuse, e.g., alcohol, cocaine, heroin, etc.), that in the Investigator's opinion may limit the subject's ability to participate or comply with study instructions and follow-up. This includes subjects with symptomatic COVID-19 infection in the past 2 months or asymptomatic COVID-19 positive test in the past 1 month.

    Angiographic Exclusion Criteria
21. Angiographic evidence of thromboembolism or atheroembolism in the target or non-target vessel as confirmed by angiography.
22. Non target lesion located in the popliteal P3 (infrageniculate) segment or treated with atherectomy.
23. Presence of aneurysm or acute thrombus in the aorta or lower extremity arteries.
24. Prior below-the-knee bypass in the target limb.
25. Previously stented lesion(s) or the presence of stents in the target vessel.
26. Target vessel(s) have distal hemodynamically significant lesions (≥ 50% diameter stenosis by angiography) outside of the allowed treatment zone (presence of non-target lesions in the target vessel is an exclusion criterion).
27. Lesions (target or non-target) with severe calcification (per PACSS 4 classification).
28. Unsuccessful treatment of stenosis (≥ 50% stenosis) of in-flow arteries including the P3 segment of the popliteal artery (infrageniculate).
29. Absence of a patent pedal artery. Absence of contiguous dorsalis pedis or common plantar arteries if the target vessels are anterior or posterior tibial arteries, respectively.
30. Target lesion location requires bifurcation treatment with scaffolding of both branches (kissing scaffold is not allowed). In case of presence of disease at a bifurcation, one vessel can be treated as target and the other as non-target.
31. Lesions (target or non-target) in which successful predilatation cannot be achieved.
32. Planned atherectomy treatment of any target or non-target lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Freedom from MALE+POD (Major Adverse Limb Event + Peri-Operative Death) | POD at 30 Days and MALE at 6 months
  Major Adverse Limb Event (MALE) includes above ankle amputation in index limb, major re-intervention on index limb at 6 months and POD includes perioperative (30-day) mortality.
Primary Efficacy Endpoint: Composite of Limb Salvage and Primary Patency | 6 months
  Composite of Limb Salvage and Primary Patency includes freedom from: above ankle amputation in index limb, 100% total occlusion of target vessel, binary restenosis of target lesion and clinically-driven target lesion revascularization (CD-TLR).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Secemsky, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Marianne Brodmann, MD, Principal Investigator — Medical University of Graz; Ramon L Varcoe, MD, Principal Investigator — Prince of Wales Private Hospital
Locations (3):
- United States (3):
  - NYU Langone Health, New York, New York
  - CUMC/NYP, New York, New York
  - Staten Island University Hospital - Northwell Health, Staten Island, New York

IPD SHARING:
Plan to Share IPD: No